CLINICAL TRIAL: NCT03957369
Title: Prevalence of NRTI, NNRTI, PI and INSTI Primary Resistance-Associated Mutations of Adult Naïve HIV-1 Seropositive Patients in Colombia
Brief Title: Primary Resistance in HIV Patients in Colombia
Status: Completed | Type: Observational
Sponsor: Fundacion REVIVA, Red de VIH del Valle del Cauca (Network)
Collaborators: ViiV Healthcare (Industry); Centro de Investigación en. Enfermedades Infecciosas, Mexico (Other Government)
Responsible Party: Sponsor
Other Study IDs: 212167
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-04

CONDITIONS: HIV Infection
Keywords: HIV infection; Primary resistance; Antiretroviral drugs; Colombia; Cross sectional study
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Collection of whole blood from study subjects from July 2021 thru July 2022, with an estimated sample size of 501 HIV positive naive individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult naive HIV positive individuals: HIV-diagnosed subjects, older than 18 years, with no prior exposure to antiretroviral drugs.
  Interventions: Diagnostic Test: HIV-1 plasma RNA Genotyping secuencing by Sanger technique; Diagnostic Test: HIV-1 plasma RNA Genotyping secuencing by Ultra-deep sequencing technique

INTERVENTIONS:
Diagnostic Test: HIV-1 plasma RNA Genotyping secuencing by Sanger technique — After signing informed consent, we will collect whole blood for HIV genotyping in plasma HIV-1 RNA for testing of resistance-associated mutations to reverse transcriptase, protease, and integrase enzymes.
  Other Names: Sanger Sequencing
Diagnostic Test: HIV-1 plasma RNA Genotyping secuencing by Ultra-deep sequencing technique — After signing informed consent, we will collect whole blood for HIV genotyping in plasma HIV-1 RNA for testing of resistance-associated mutations to reverse transcriptase, protease, and integrase enzymes.
  Other Names: Next-Generation Sequencing

SUMMARY:
The investigators' main objective is to determine the prevalence of pre-treatment of resistance-associated mutations (RAMs) in a naïve and recently diagnosed HIV infection in 18 centers from 12 cities in Colombia. This evaluation will include the genotyping of all three enzymes, reverse transcriptase, protease, and integrase. This type of complete primary resistance profile has not yet been reported in Colombia and there is only scanty data regarding resistance-associated mutations to NRTIs, NNRTIs, and PIs in the country

DETAILED DESCRIPTION:
The number of patients and sample size:

The proportion formula for finite populations was used to determine the sample size (with appropriate confidence intervals) needed to find the prevalence of RAMs in naive HIV population from Colombia.

As shown below, estimating 20% of loss, the sample size will be 500 study subjects considering a CI 97%.

The sample size is estimated in 501 patients, considering 1% or less of the probability of finding pre-treatment resistance-associated mutations affecting integrase inhibitors, a CI of 97%, and 20% of blood samples loss or not processable.

Sample selection:

The investigators chose 12 cities (Bogotá, Cali, Medellín, Barranquilla, Montería, Cartagena, Bucaramanga, Cúcuta, Pereira, Villavicencio, Pasto, and Florencia) in which the majority of the HIV population is found in Colombia, accounting for around 80% according to data from the High-Cost Account (CAC, in its Spanish acronym) 2016. Moreover, this allows the selection of patients with diverse races or ethnic groups.

The healthcare provider institutions (Instituciones Prestadoras de Salud - IPS in Spanish) with integral HIV care programs in accordance with the quality and service requirements demanded by the Colombian Ministry of Social Protection.

The sample will be selected as follows:

1. Patients will be chosen based on the opportunity to attend the healthcare provider institutions (IPS) if they meet the inclusion criteria.
2. Treating physicians in charge of HIV care in the healthcare provider institutions will invite patients to participate upon explanation of the nature, purposes, and benefits of the study. If a patient agrees to participate, informed consent will be asked. Once this consent is given and the respective written form is signed, the collection of data will be collected and a blood sample will be drawn.
3. If a patient has signed the written informed consent form but does not provide the blood sample, he or she will be excluded and another patient will be expected to be included in order to complete the sample size calculated for the study.

Data collection:

A unique identification code, assigned to each patient, will be registered in the case report forms and in the laboratory report. The research group will keep the absolute privacy of collected data that relates the patient's name with the identification code.

Procedures for primary resistance-associated mutations determination in the blood samples:

Genotyping sequencing will be performed using traditional and ultradeep sequencing techniques in plasma samples by Sanger and Next-Generation Sequencing, respectively. Stanford database analysis criteria will be used to compare the performance of these techniques. Both techniques will be performed in all samples.

Plasma samples will be sent for processing for both techniques at Centro de Investigación en Enfermedades Infecciosas - CIENI in Mexico City.

ELIGIBILITY:
Inclusion Criteria:

1. Naive HIV-positive individuals aged 18 years or older.
2. Consent to participate in the research.

Exclusion Criteria:

1. Patients with any type of antiretroviral exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with HIV infection not exposed to any HIV antiretroviral drugs, regardless of the time of the HIV diagnosis
Sampling Method: Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of primary HIV drug associated resistance in Colombia | November 2019 - December 2020
  Prevalence estimated by nationwide sampling of adults HIV positive individuals

SECONDARY OUTCOMES:
Outcomes by demographic characteristics | November 2019 - September 2022
  Estimate HIV drug resistance by age, sex, race and ethnic groups overall and in each of the different included Colombian regions and 12 Colombian cities
Resistance to integrase | November 2019 - September 2022
  Determine the presence of RAMs to integrase to correlate with primary resistance to integrase inhibitors in Colombia
Correlate of HIV-1 sequencing by Sanger vs Next-Generation Sequencing techniques | November 2019 - September 2022
  Compare the results from sequencing plasma HIV-1 RNA by both proposed techniques

CONTACTS AND LOCATIONS:
Overall Officials: ERNESTO MARTINEZ, Principal Investigator — Fundacion REVIVA, Red de VIH del Valle del Cauca
Locations (1):
- REVIVA, Red de VIH del Valle del Cauca, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No